CLINICAL TRIAL: NCT01949103
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose (MAD) Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TD-1607, a Glycopeptide-Cephalosporin Heterodimer Antibiotic, in Healthy Subjects
Brief Title: TD-1607 MAD Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0104
Record Dates: First submitted 2013-09-17; First posted 2013-09-24 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Infections; Bacterial Infections
Keywords: Gram-positive
MeSH Terms: conditions — Infections; Bacterial Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- TD-1607 or placebo (Dose1) (Experimental): TD-1607 or placebo administered intravenously
  Interventions: Drug: TD-1607; Drug: Placebo
- TD-1607 or placebo (Dose 2) (Experimental): TD-1607 or placebo administered intravenously
  Interventions: Drug: TD-1607; Drug: Placebo
- TD-1607 or placebo (Dose 3) (Experimental): TD-1607 or placebo administered intravenously
  Interventions: Drug: TD-1607; Drug: Placebo
- TD-1607 or placebo (Dose 4) (Experimental): TD-1607 or placebo administered intravenously
  Interventions: Drug: TD-1607; Drug: Placebo
- TD-1607 or placebo (Dose 5) [Optional] (Experimental): TD-1607 or placebo administered intravenously
  Interventions: Drug: TD-1607; Drug: Placebo
- TD-1607 or placebo (Dose 6) [Optional] (Experimental): TD-1607 or placebo administered intravenously
  Interventions: Drug: TD-1607; Drug: Placebo

INTERVENTIONS:
Drug: TD-1607
Drug: Placebo

SUMMARY:
TD-1607, administered intravenously as multiple ascending doses, will be investigated in healthy subjects to assess its tolerability, safety, and pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy nonsmoking male or a female (of non-childbearing potential) and 18 to 55 years old, inclusive, at Screening.
* Subject has a body mass index (BMI) of 19 to 30 kg/m2, inclusive, and weighs at least 50 kg.

Subject has no clinically significant abnormalities in the results of laboratory evaluations at Screening and Day -1.

Exclusion Criteria:

* Subject has evidence or history of clinically significant, relevant hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (except for untreated, asymptomatic seasonal allergies at time of dosing).
* Subject has a history of allergies or hypersensitivities to glycopeptide (e.g., vancomycin) or beta-lactam (e.g., penicillin or cephalosporin) antibiotics.
* Subject has participated in another clinical trial of an investigational drug (or medical device) within 60 days (or 5 half-lives, whichever is longer) prior to Screening or is currently participating in another trial of an investigational drug (or medical device).
* Subject has previously participated in a trial for TD-1607.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 17 days
  Adverse events

SECONDARY OUTCOMES:
Cmax | 17 Days
  Pharmacokinetics
Tmax | 17 Days
  Pharmacokinetics
AUC0-t | 17 Days
  Pharmacokinetics
AUC0-24 | 17 Days
  Pharmacokinetics
AUCinf | 17 Days
  Pharmacokinetics
CL | 17 Days
  Pharmacokinetics
Vdss | 17 Days
  Pharmacokinetics
t1/2 | 17 Days
  Pharmacokinetics
Amount excreted in urine (Ae | 17 Days
  Pharmacokinetics
Fraction eliminated in urine (fe) | 17 Days
  Pharmacokinetics
CLr | 17 Days
  Pharmacokinetics
Ctrough | 17 Days
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- PPD, Phase 1 Clinic, Austin, Texas, United States